CLINICAL TRIAL: NCT00418600
Title: A Phase 4, Multi-Center, Open-Label, Randomized Study to Determine Clinically Appropriate Doses of Hectorol® Capsules When Converting From Hectorol® Injection for the Treatment of SHPT in Stage 5 CKD Subjects on Hemodialysis
Brief Title: A Phase 4, Conversion Study of Hectorol® Injection to Hectorol® Capsules in Stage 5 CKD Patients on Dialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HECT00406
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Secondary Hyperparathyroidism; Hectorol® (doxercalciferol capsules); Hectorol® (doxercalciferol injection)
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — 1 alpha-hydroxyergocalciferol

ARMS (3):
- 1 (Other): Hectorol capsules at 1.0 times current injection dose
  Interventions: Drug: Hectorol® (doxercalciferol capsules)
- 2 (Other): Hectorol capsules at 1.5 times current injection dose
  Interventions: Drug: doxercalciferol capsules, Hectorol®
- 3 (Other): Hectorol capsules at 2.0 times current injection dose
  Interventions: Drug: doxercalciferol capsules, Hectorol® capsules

INTERVENTIONS:
Drug: Hectorol® (doxercalciferol capsules) — Hectorol capsules at 1.0 times current injection dose
  Arms: 1
Drug: doxercalciferol capsules, Hectorol® — Hectorol capsules at 1.5 times current injection dose
  Arms: 2
Drug: doxercalciferol capsules, Hectorol® capsules — Hectorol capsules at 2.0 times current injection dose
  Arms: 3

SUMMARY:
Hectorol is a safe and effective treatment of secondary hyperparathyroidism in hemodialysis patients. Hectorol (doxercalciferol capsules) is indicated for the treatment of secondary hyperparathyroidism in patients with chronic kidney disease on dialysis and in pre-dialysis patients with Stage 3 or Stage 4 chronic kidney disease. Hectorol (doxercalciferol injection) is indicated for the treatment of secondary hyperparathyroidism in patients with chronic kidney disease on dialysis.

This protocol will determine clinically appropriate doses of Hectorol (doxercalciferol capsules) when converting subject from Hectorol (doxercalciferol injection.) The study will enroll hemodialysis patients that have been controlled on intravenous Hectorol. the information gained from this study will be a useful guide for physicians in managing CKD Stage 5 patients for whom a change from intravenous to oral vitamin D administration is appropriate.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be receiving hemodialysis three times per week for a minimum of six months.
* The subject must have been receiving Hectorol Injection for a minimum of 3 months. The subject must have been on a stable dose regimen, three times per week administration for a minimum of four weeks.
* The central laboratory assessment must be within the following ranges: serum iPTH between 150-600 pg/mL, inclusive; corrected calcium < 10.0 mg/dL; phosphorus < 7.0 mg/dL.

Exclusion Criteria:

* In the opinion of the Investigator, the subject currently has poorly controlled diabetes mellitus, poorly controlled hypertension, active vasculitis, HIV infection, or any other clinically significant, unstable medical condition.
* Abnormal liver function as measured by ALT/AST greater than two times the upper limit of normal (ULN).
* The subject currently has malabsorption, severe chronic diarrhea, or ileostomy.
* Any evidence of active malignancy except for basal cell carcinoma of the skin. A history of malignancy is not an exclusion.
* Current use of aluminum or magnesium based binders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-11; Primary Completion 2007-06 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Dose Conversion | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (8):
  - Hot Springs, Arkansas
  - Downey, California
  - Tarzana, California
  - Atlanta, Georgia
  - Cincinnati, Ohio
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Spokane, Washington

REFERENCES:
- See also: US FDA Approved Full Prescribing Information for Hectorol® Capsules — http://www.hectorol.com/docs/Hectorol%20Capsule%20PI%20Text_2006-01.pdf
- See also: US FDA Approved Full Prescribing Information for Hectorol® Injection — http://www.hectorol.com/docs/Hectorol%20Injection%20PI%20Text_2006-01.pdf